CLINICAL TRIAL: NCT06584968
Title: Improving the Application Skill of Semmes-Weinstein Monofilament Test with Different Teaching Methods: a Randomized Controlled Trial
Brief Title: Improving the Application Skill of the Semmes-Weinstein Monofilament Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Ozge Buket Arslan, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SWMTeaching
Record Dates: First submitted 2024-08-21; First posted 2024-09-05 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Training; Students
MeSH Terms: interventions — Feedback, Sensory

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training with visual feedback (Experimental): The students in the study group will do monofilament applications on a precision scale. They will be provided with visual feedback by comparing the value of the monofilament with the pressure value of the monofilament applied on the precision scale in grams. In this way, the students will visually experience whether they can provide the appropriate level of pressure during the application. The practice on the precision scale will continue for 15-20 minutes with the monofilaments in the Semmes-Weinstein Monofilament Test kit.
  Interventions: Other: training with visual feedback
- Classical learning (Active Comparator): The students in the control group will do practical applications with the classical learning method, where one of the researchers plays the patient role. They will do application trials with the monofilaments in the Semmes-Weinstein Monofilament Test kit for 15-20 minutes.
  Interventions: Other: classical learning

INTERVENTIONS:
Other: training with visual feedback — Training with visual feedback by comparing the value of the monofilament with the pressure value of the monofilament applied on the precision scale in grams.
  Arms: Training with visual feedback
Other: classical learning — Study of the test with practical applications on the researcher who plays the role of the patient
  Arms: Classical learning

SUMMARY:
The Semmes-Weinstein Monofilament Test is one of the most widely used and objective clinical tests for assessing the sense of touch. Some guides include standard instructions for the application of the Semmes-Weinstein Monofilament Test. With monofilaments applied correctly by the instructions, patients' threshold values can be determined accurately. However, there are disagreements about the accuracy of the pressure applied by the therapist who applies the monofilament to the patient. The investigators aimed to compare the application of the Semmes-Weinstein Monofilament Test to undergraduate students of the occupational therapy department by teaching it using classical methods and visual feedback.

ELIGIBILITY:
Inclusion Criteria:

* Being third or fourth-year undergraduate students of the Occupational Therapy Department
* Completing the Hand Rehabilitation course
* Being a volunteer to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Application duration of the Semmes-Weinstein Monofilament Test | just before the intervention and just after completion of the intervention
  The application duration of the Semmes-Weinstein Monofilament Test will be recorded in seconds.
The applied force of the Semmes-Weinstein Monofilament Test | just before the intervention and just after completion of the intervention
  The applied force of the Semmes-Weinstein Monofilament Test will be recorded in grams.
Intervals between the Semmes-Weinstein Monofilament Test applications | just before the intervention and just after completion of the intervention
  Intervals between the Semmes-Weinstein Monofilament Test applications will be recorded in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided